CLINICAL TRIAL: NCT06255418
Title: Big Data and Real-world Evidence to Assess the Healthcare and Health Outcomes Burden of Acute Coronary Syndromes Complicated With Heart Failure: the BEAT-HF Study
Brief Title: Big Data to Assess the Healthcare and Health Outcomes Burden of Acute Coronary Syndromes Complicated With Heart Failure
Acronym: BEAT-HF
Status: Completed | Type: Observational
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Institut d'Investigació Biomèdica de Bellvitge (Other)
Responsible Party: Principal Investigator, Josep Comín, Director of Innovation, Research and Universities of the South-Metropolitan Healthcare Area, Hospital Universitari de Bellvitge
Other Study IDs: PR251/22
Record Dates: First submitted 2024-02-04; First posted 2024-02-13 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure; Acute Coronary Syndrome; Heart Decompensation; Myocardial Infarction, Acute
Keywords: heart failure; acute coronary syndrome; real-world evidence; healthcare resources consumption; long-term heart failure; big data
MeSH Terms: conditions — Heart Failure; Acute Coronary Syndrome; Myocardial Infarction

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to define the incidence of heart failure (HF) after acute coronary syndrome (ACS). The main question it aims to answer is:

• To define HF incidence in the medium and long-term in the context of public healthcare coverage ensuring universal access to early coronary revascularization after ACS and extended neurohormonal treatment.

Analyses will cover the entire population of Catalonia (North-Eastern region of Spain, N = 7.860.563 in 2020).

Researchers will compare HF incidence rate according to relevant subgroup characteristics including event type, age groups or sex, inter alia.

DETAILED DESCRIPTION:
The aim of this project is to gain a better understanding, from a population perspective, of incident heart failure (HF) after acute coronary syndrome (ACS). The particular purpose is to define its incidence in the medium and long-term in the context of public healthcare coverage ensuring universal access to early coronary revascularization after ACS and extended neurohormonal treatment. To provide answer to this objective, a retrospective study were designed where a variety of study designs and analytic approaches will be used, aimed at maximizing the robustness of the results and at minimizing their sensitivity to specific study design assumptions. Analyses will cover the entire population of Catalonia (Spain, N = 7.860.563 as of December 31st, 2020), a region in which the Catalan Health Service granted universal health coverage. The study period will be defined between January 1st, 2012, and December 31st, 2021 covering 10 years. Inclusion criteria will be to have been admitted and diagnosed with a primary diagnosis of ACS (non-ST-segment elevation myocardial infarction -NSTEMI-, ST-segment elevation myocardial infarction -STEMI-, unstable angina -UA-) during the index event and to have been discharged alive during this period. The first co-primary outcome is to define the baseline characteristics of the ACS population, overall and according to clinical interest groups including event type (STEMI, NSTEMI, UA) and other relevant subgroups of patients. The second co-primary outcome of the study is the incidence rate of HF after ACS of all patients discharged alive after an ACS in Catalonia during this period. Incidence rate will also be described overall and according to relevant subgroup characteristics including event type, clinical phenotypes surrogate of impairment in regional or global systolic function, age groups, sex, diabetes mellitus, HF complicating index ACS, recurrent ACS after index ACS, socioeconomic status, treatments, comorbidity groups and procedures. Other clinical outcomes will be assessed as secondary outcomes (all-cause death, stroke, recurrent ACS, hospitalizations, major adverse cardiac event, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Admission with the primary diagnosis of acute coronary syndrome ( Non-ST-Elevation Myocardial Infarction -NSTEMI-, ST-Elevation Myocardial Infarction -STEMI-, Unestable Angina -UA-)

Exclusion Criteria:

* Diagnosis of heart failure (HF) in the year preceding the inclusion.
* Death before discharge from index event.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Analyses will cover the entire population of Catalonia (Spain, N = 7.860.563 as of December 31st, 2020), a region in which the Catalan Health Service granted universal health coverage.
Sampling Method: Non-Probability Sample
Enrollment: 7860560 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Baseline characteristics | Between January 1st, 2012 and 31st, December 2021 (study period).
  The first co-primary outcome is to define the baseline characteristics of the ACS population, overall and according to clinical interest groups including event type (STEMI, NSTEMI, UA) and other relevant subgroups of patients.
Incidence of heart failure after acute coronary syndrome | Between January 1st, 2012 and 31st, December 2021 (study period).
  The second co-primary outcome of the study is the incidence rate of HF after ACS of all patients discharged alive after an ACS in Catalonia

SECONDARY OUTCOMES:
Clinical endpoints | Between January 1st, 2012 and 31st, December 2021 (study period).
  * All-cause death
  * Left ventricular assist device (LVAD) implant
  * Heart transplant (HTx)
  * Need of cardiovascular (CV) procedures: coronary artery bypass grafting (CABG), percutaneous revascularization, implantable cardioverter-defibrillator (ICD) implant
  * Recurrent acute coronary syndromes (ACS)
  * Stroke
  * Cardiovascular (CV)-related hospitalization
  * Heart Failure (HF) hospitalization
  * 5-point MACE: death, incident HF, new ACS, stroke, need of cardiovascular intervention (CABG or percutaneous revascularization)
  * Relevant cardiovascular medication by therapeutic class during the first year after the event.
Healthcare resource use endpoints | Between January 1st, 2012 and 31st, December 2021 (study period).
  * Emergency Department (ED) visits
  * Daycare visits
  * Outpatient specialist contacts
  * Total primary care contacts
  * Primary care nurse contacts
  * Primary care physician contacts
  * Use of skilled nurse facility
  * Unplanned HF admission
  * Unplanned CV readmission
  * Unplanned clinically related readmission (includes CV readmissions, admissions related to pre-existing chronic non-CV conditions and complications attributable to the index hospitalization)
  * Unplanned all-cause hospitalization
  * Length of hospitalization (days per admission)
  * Healthcare expenditure: global and stratified according to specific concepts and activities
  * Drug costs

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain